CLINICAL TRIAL: NCT03994185
Title: Prospective Investigation of The Merit WRAPSODY™ Endovascular Stent Graft for Treatment of Iliac Artery Occlusive Disease
Brief Title: The Merit WRAPSODY™ Endovascular Stent Graft for Treatment of Iliac Artery Occlusive Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was withdrawn by the Sponsor prior to enrollment
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IOD-P2-19-01
Record Dates: First submitted 2019-06-19; First posted 2019-06-21 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Stenosis of Artery; Peripheral Arterial Disease; Iliac Artery Disease; Iliac Artery Occlusion
Keywords: PAOD; Peripheral Arterial Occlusive Disease; Iliac Artery Disease; Stent Graft
MeSH Terms: conditions — Peripheral Arterial Disease; Peripheral Arterial Occlusive Disease 1

STUDY DESIGN:
Intervention Model Description: Approximately 30 subjects will be enrolled and treated with the study device
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Group Treated with stent graft (Experimental): This is a single arm study. All subjects will be treated with the WRAPSODY stent graft.
  Interventions: Device: Placement of WRAPSODY stent graft

INTERVENTIONS:
Device: Placement of WRAPSODY stent graft — Placement of WRAPSODY stent graft into the iliac arteries and/or aortic bifurcation.

SUMMARY:
This is a prospective, single-center, non-randomized phase 2, first-in-iliac artery study, to evaluate the safety and effectiveness of the WRAPSODY Stent Graft for the treatment of peripheral arterial occlusive disease in symptomatic subjects with de novo or restenotic lesions in the common iliac artery (CIA) and/or external iliac artery (EIA), including lesions at the aortic bifurcation.

DETAILED DESCRIPTION:
Approximately 30 subjects will be enrolled. Post study procedure subjects will have planned follow-up visits at 4 weeks, 24, 36 and 52 weeks, and unscheduled visits as medically necessary,

The primary study safety endpoint is the proportion of subjects free from a composite of device- or procedure-related death, myocardial infarction, or amputation above the metatarsals in the treated leg resulting from a vascular event, or device- or procedure-related serious adverse events within 4 weeks of the index procedure. The primary clinical effectiveness endpoint is the proportion of subjects with a composite improvement of at least 1 Rutherford category and patency as evaluated by duplex ultrasound at 4 weeks after index procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has signed informed consent
2. Subject is ≥ 21 years of age
3. Subject is able and willing to comply with study requirements
4. Male, infertile female, or female practicing contraception and a negative pregnancy test within 7 days prior to the study procedure
5. Symptomatic claudication or rest pain without tissue loss, Rutherford category 2-4
6. Angiographic evidence of de novo or restenotic target lesion(s) in native vessels in the common and/or external iliac artery(ies) (multiple stenoses may exist within the target lesion)
7. Total lesion(s) length is ≤ 110mm
8. Target lesion(s) is at least 3 cm from an existing stent or stent graft
9. At least 1 stenosis in the target vessel has ≥ 50% stenosis
10. Target vessel diameter is between 4.6 and 14.4mm at angiographic screening for device placement
11. Adequate ipsilateral blood flow, including at least 1 patent (<50% stenotic) superficial femoral or profundal femoral artery
12. Full expansion of an appropriately sized (in the investigator's opinion) standard angioplasty balloon has been achieved during primary angioplasty at the target lesion prior to enrollment

Exclusion Criteria:

1. Subject has undergone an intervention (surgical or percutaneous) in the target limb(s) <30 days from the date of the index study procedure
2. Subject has a surgical or percutaneous procedure in the target limb(s) planned within 30 days following the index study procedure
3. Previous or planned bypass surgery in the target limb(s)
4. Coronary intervention within 30 days prior to enrollment or planned within 12 months after index study procedure
5. Subject has had a stroke within 90 days prior to the index study procedure
6. Subject has had a transient ischemic attack within 30 days prior to the index study procedure
7. Uncorrectable coagulation disorder
8. Subject cannot receive heparin, dual antiplatelet treatment, or anticoagulant(s) appropriate in the opinion of the investigator
9. Condition unrelated to study anticipated to require indefinite anticoagulation
10. Evidence of blood borne infection
11. Hypersensitivity to nickel titanium alloy
12. Allergy to radiographic contrast material which cannot be adequately premedicated
13. Serum creatinine >2.5mg/dL
14. The subject is enrolled in another investigational study
15. Life expectancy is ≤ 12 months
16. Active malignancy other than non-melanomatous skin cancer
17. Stenosis/restenosis is located within a previously placed stent or stent graft
18. Angiographic evidence of thrombus within or adjacent to the target lesion(s)
19. Aneurysmal dilation proximal or distal to the target lesion(s) that could interfere with placement of the study device
20. Abdominal aortic artery stent, if it could interfere with placement of the study device
21. Target lesion(s) are located such that the stent graft would prevent blood flow to the internal iliac artery, if patent
22. Lesions requiring atherectomy or ablation to facilitate stent graft delivery
23. Any other condition deemed exclusionary in the opinion of the investigator for documented reasons relating to the health and/or welfare of the subject

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2020-09 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety endpoint of subjects free from specified adverse events | 4 weeks after placement of WRAPSODY stent graft
  The primary study safety endpoint is the proportion of subjects free from a composite of device- or procedure-related death, myocardial infarction, or amputation above the metatarsals in the treated leg resulting from a vascular event, or device- or procedure-related serious adverse events within 4 weeks of the index procedure.
Effectiveness endpoint of subjects with improvement of Rutherford Category | 4 weeks after placement of WRAPSODY stent graft
  The primary clinical effectiveness endpoint is the proportion of subjects with improvement of at least 1 Rutherford category within 4 weeks of the index procedure. Composite with Outcome 3.
Effectiveness endpoint of subjects with patency | 4 weeks after placement of WRAPSODY stent graft
  The primary clinical effectiveness endpoint is the proportion of subjects with patency as evaluated by duplex ultrasound at 4 weeks after index procedure. Composite with Outcome 2.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Holden, Principal Investigator — Auckland City Hospital

IPD SHARING:
Plan to Share IPD: No